CLINICAL TRIAL: NCT04155762
Title: A Comparison of the Effects of Pin and Vacuum Assisted Suspension Systems in Transtibial Amputees
Brief Title: Effects of Pin and Vacuum Assisted Suspension Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Senay Cerezci Duygu, Research Assistant, Baskent University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GO 15/123
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Amputees; Prosthesis User; Artificial Limbs
Keywords: Amputees; Artificial Limbs; Prosthetic designs; Rehabilitation of prostheses users; Prosthetic suspension systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Both suspension systems were applied consecutively to the participants. Initially, participants used the Pin Suspension System (PSS) for three months following fabrication and adjustment of the prosthesis, and a prosthetic training period. They then employed the Vacuum-Assisted Suspension System (VASS) for three months after a similar training period.
  Interventions: Other: Pin Suspension System (a prosthetic suspension system); Other: Vacuum-Assisted Suspension System (a prosthetic suspension system)

INTERVENTIONS:
Other: Pin Suspension System (a prosthetic suspension system) — Participants used the PSS for three months following fabrication and adjustment of the prosthesis, and a prosthetic training period.
Other: Vacuum-Assisted Suspension System (a prosthetic suspension system) — After PSS, participants employed the VASS for three months after a similar training period.

SUMMARY:
This study was performed to determine the presence of any difference between Pin Suspension (PS) and Active Vacuum Suspension (AVS) on walking capacity, functional mobility, weight bearing in the prosthetic side, prosthetic satisfaction and body image were evaluated. Nine patients who don't have an obstacle to both socket applications in terms of stump height, type and edema were evaluated in this study. Both suspension systems were administered to the patients included in the study. First, amputees have used PS for 3 months following alignment of the prosthesis and training period. Then again they used AVS for 3 months following alignment of the prosthesis and training period. For each system, after adapting prosthesis 'LASAR posture' was used to evaluate weight bearing on the prosthetic side, '6 Minute Walk Test' for walking capacity, 'Time Up and Go' test for functional mobility, 'Prosthetic Satisfaction Index' for prosthetic satisfaction and 'Amputee Body Image Scale' for body. There were statistically significant difference between PS and AVS in terms of prosthetic side weight bearing percentage, walking capacity, functional mobility and prosthetic satisfaction (p<0.05), in favor of AVS. There were not statistically significant difference between the body image scores (p>0.05). From the view of function and prosthetic satisfaction, AVS was found to be more effective in transtibial amputees. It is believed that our study will be a guide to the future studies including higher number of amputees, different amputation levels and different suspension systems.

ELIGIBILITY:
Inclusion Criteria:

* Being able to walk without the use of any assistive device,
* Having normal range of motion in the hip and knee at the amputated side.

Exclusion Criteria:

* Having any disadvantage about prosthetic device usage in terms of stump length, shape and edema,
* Having movement limitation,
* Having any discomfort or health problem (cardiopulmonary, neurological or orthopedic problems) that may affect gait other than amputation,
* Having multiple extremity loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Weight-bearing on the prosthetic side | 3 minutes
  The percentage of total body weight borne on the amputated limb will be recorded.
Walking capacity | 6 minutes
  "Six Minutes Walk Test" will be used to assess walking capacity. Participants will walk for 6 minutes between two points which are 24 meters apart. The total meters walked during those 6 minutes will be recorded.
Functional mobility | 1 minute
  "The Timed Up and Go Test" will be used to assess functional mobility. The test starts from the seated position on the chair. With the onset of time, the participant leaves the chair, walks for 3 meters, turns 180 degrees, returns to the starting point, and sits in the chair back. The test is finished when the participant is returned to the initial position and the total time is recorded in seconds.
Prosthetic satisfaction | 5 minutes
  "Satisfaction with Prosthesis Questionnaire" (SAT-PRO) is a self-administered questionnaire for determining the participants' satisfaction with the use of the prosthesis. It consists of 15 items. For each item, participants mark the number that best describes their satisfaction with current prosthesis (3: totally agree, 2: rather agree, 1: rather disagree, 0: totally disagree). The items 6, 12 and 14 are scored in reverse. In total, lower scores indicate higher satisfaction; the maximum score that can be taken in the questionnaire is 45 points which means 100% satisfaction and 0 points means 0% satisfaction.
  The Turkish version of the SAT-PRO is a valid and reliable test that can be used to evaluate the prosthetic satisfaction of people with lower extremity amputation.
Body image perception | 5 minutes
  "The Amputee Body Image Scale" (ABIS) is a self-administered questionnaire for determining how an amputee perceives and feels about his/her body experience. It consists of 20 items. The items 3, 12 and 16 are scored in reverse. The total score varies from 20 to 100; lower scores indicate better body image.
  The Turkish version of the ABIS was found to be valid and reliable.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Erbahceci, Prof, Study Chair — Hacettepe University; Bahar Kulunkoglu, Assoc Prof, Principal Investigator — Ankara Yildirim Beyazıt University; Senay Cerezci Duygu, MsC, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No